CLINICAL TRIAL: NCT04664114
Title: The Effect of Viewing Images of Fetus to Pregnant Women With Virtual Reality Glasses on Birth Pain, Perception and Anxiety During Labor
Brief Title: The Effect of Virtual Reality Glass During Labor Process on Labor Pain, Birth Perception and Anxiety
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mine Yilmaz Koçak, Lecturer, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/259
Record Dates: First submitted 2020-11-10; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Birth, First
Keywords: birth; Virtual reality; anxiety; pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled experimental study. The study intervention group was carried out with a total of 100 pregnant women, 50 of whom were controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Both the evaluation of the fetus and the ultrasound for visual purposes took 15-20 minutes in total. These pregnant women were asked to bring their mobile phones with them during delivery. When the birth of the pregnant woman started, she was hospitalized by the third researcher. The follow-up and deliveries during the labor were carried out by the 3rd and 4th researchers. With an application installed on the pregnant woman's phone, these two-dimensional images were transformed into three-dimensional images and the pregnant women were watched consecutively with the VR Box 3D virtual reality glasses. In cases where the program was not compatible with the phone of the pregnant woman, the researcher was watched by the midwife. The total image viewing time was recorded.
  Interventions: Behavioral: Virtual Reality
- Control Group (No Intervention): Only one pregnant woman was included in the study at the same time in order to avoid any interruption in the follow-up of the pregnant women. VAS was applied to women in both groups when cervical dilatation was 4 and 9 cm. Approximately two hours after giving birth (to allow mothers to breastfeed their babies and to stabilize the mother's vital signs), the Women's Perception of Supportive Care at Birth Scale and the Perinatal Anxiety Screening Scale were applied.

INTERVENTIONS:
Behavioral: Virtual Reality — Ultrasound images of the fetus in the 28th week of pregnancy of the women in the intervention group were recorded. These images were shown to the woman through virtual reality glasses during the labor. Routine practices in the hospital were made to the women in the control group. VAS (Visual Analog Scale) was applied to women in both groups when cervical dilatation was 4 and 9 cm. Approximately two hours after giving birth (to allow mothers to breastfeed their babies and to stabilize the mother's vital signs), the Women's Perception of Supportive Care at Birth Scale (POBS) and Perinatal Anxiety Screening Scale (PASS) were administered.
  Other Names: Ultrasonography (USG)
  Arms: Experimental group

SUMMARY:
Aim: This study was conducted to determine the effect of showing images of the fetus to the pregnant women with the virtual reality glass during labor process on labor pain, birth perception and anxiety level.

Background: Virtual reality (VR) is an effective and inexpensive method that allows the creation of simulated scenarios in which it interacts with the virtual environment with multisensory stimuli.

Methods: This is a randomized controlled experimental study. The study included 100 pregnant women of whom 50 in the intervention group and 50 in the control group. Ultrasound images of the fetus were recorded on the 28th week of pregnancy of the women in the intervention group. These images were shown to the women with the virtual reality glass during labor process. Routine procedures were carried out for the women in the control group. The Visual Analog Scale (VAS) was applied to both groups when cervical dilatation was 4 cm and 9 cm. The Women's Perception for the Scale of Supportive Care Given During Labor (POBS) and the Perinatal Anxiety Screening Scale (PASS) were applied almost two hours after labor.

Keywords: Virtual reality, labor, pain, anxiety.

DETAILED DESCRIPTION:
Performed on the pregnant women in the intervention group (Virtual Reality Glass Group-VRGG) Pregnant women who met the inclusion criteria and were in the 28th weeks of pregnancy were assigned in the intervention or control group according to the randomization chart when they came to the Obstetrics and Gynecology Polyclinic for pregnancy follow-up. Pregnant women in the intervention group were informed about the study, and their verbal and written consent was obtained. The third author and the Gynecology and Obstetrics Specialist evaluated the presentation of the baby, amniotic fluid, placenta, umbilical artery doppler, fetal biometry (BPD, HC, AC, FL) and fetal respiration with the Voluson 730 PRO ultrasound device. In the remaining time, if the position of the baby is suitable, it was ensured that video images were recorded on the phone of the pregnant woman by looking at the baby's face with the help of a 3D / 4D probe. Although it might be performed in earlier and later weeks, such visual evaluations are made in the 27th-28th weeks since the visualization is better. The ultrasound session both for the evaluation of the fetus and for visual purposes took 15-20 minutes in total. These pregnant women were asked to bring their phone that the video was recorded with them to the labor. When the pregnant women got into labor, they were hospitalized by the third researcher. The follow-ups and labor were also performed by the third author. These two-dimensional images were converted into three-dimensional images through an application installed in the mother's phone and were shown to her with a VR Box 3 D virtual reality glass one after another. In cases where the program was not compatible with the mother's phone, it was watched on the researcher's phone. The total duration of image viewing was recorded.

Practices performed on the pregnant women in the control group (Control Group-CG) Pregnant women who met the inclusion criteria and were in the 28th weeks of pregnancy were assigned to the control group according to the randomization chart. When the pregnant women got into labor, they were hospitalized by the third researcher. No practices other than the routine were applied on pregnant women in the control group. These routine practices are monitoring pregnant women's cervical dilation, contraction and fetal heart rate, providing freedom of action, restricting oral intake for labor duration. No oxytocin induction or any analgesic were applied on the pregnant women in both groups. The rooms where the pregnant women stayed were kept dim and calm. The pregnant women in the control group were monitored and delivered by the third author during the labor process. For not hampering the monitoring of pregnant women, only one pregnant woman was included in the study at the same time. The Visual Analog Scale (VAS) was applied to both groups when cervical dilatation was 4 cm and 9 cm. The Women's Perception for the Scale of Supportive Care Given During Labor (POBS) and the Perinatal Anxiety Screening Scale (PASS) were applied almost two hours after labor (so that the mother had time to breastfeed the baby and the mother's vital signs were stabilized).

ELIGIBILITY:
Inclusion Criteria:

* at 28 weeks of gestation (because the images of the fetus can be taken more clearly)
* Primipara,
* Having a head presentation,
* Without any risk conditions related to the pregnant and fetus (preeclampsia, gestational diabetes, presentation anomalies, placenta related anomalies, fetal distress and anomaly),
* Over the age of 18,
* Can understand and speak Turkish,
* Pregnant women who agreed to participate in the study after giving information about the study

Exclusion Criteria:

* Elective cesarean section
* Conceived with assisted reproductive techniques
* Pregnant women with vision and hearing problems were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregmant women
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The progression time of vaginal dilatation at birth may vary from person to person. For this reason, measurement will be made when the vaginal dilatation is 4 cm from the beginning of the birth process.
  Birth pain. VAS is a horizontal or vertical line of 10 cm/100 mm that starts with "No pain" and ends with "Unbearable pain." No pain is written on one end and very severe or unbearable pain is written on the other end on the scale during the measurement and the patient marks their current state on this line. The length of the distance from no pain to the point marked by the patient indicates the patient's pain.
Visual Analog Scale (VAS) | The progression time of vaginal dilatation at birth may vary from person to person. For this reason, measurement will be made when the vaginal dilatation is 9 cm from the beginning of the birth process.
  Birth pain. VAS is a horizontal or vertical line of 10 cm/100 mm that starts with "No pain" and ends with "Unbearable pain." No pain is written on one end and very severe or unbearable pain is written on the other end on the scale during the measurement and the patient marks their current state on this line. The length of the distance from no pain to the point marked by the patient indicates the patient's pain.
Perinatal Anxiety Screening Scale (PASS) | Birth time can vary from person to person. For this reason, measurement will be made when it is 2 hours after the end of labor.
  women's anxiety level.The Perinatal Anxiety Scale (PASS) has 31 items. It is a valid and reliable scale that can be used to screen anxiety disorders among perinatal women. The answers to the questions in the scale are "never," "sometimes," "often" and "almost always" and the scores are 0, 1, 2, 3 and its cutoff score is 16.
Perception for the Scale of Supportive Care Given During Labor (POBS) | Birth time can vary from person to person. For this reason, measurement will be made when it is 2 hours after the end of labor.
  women's birth perception level. The Perception for the Scale of Supportive Care Given During Labor (POBS) scale has 33 items. It was determined to be valid and reliable to measure the women's perception for the supportive care given during labor. It is recommended to use within the first 24 hours after labor. The scale has three subdimensions. The first dimension includes behaviors that make women feel comfortable, the second dimension includes informative behaviors and the third dimension includes behaviors that disturb women. The lowest possible score obtained from the scale is 33 while the highest score is 132. It has no cut-off point. Higher scores indicate well-perceived supportive care.

CONTACTS AND LOCATIONS:
Locations (1):
- Mine Yilmaz Koçak, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akin B, Yilmaz Kocak M, Kucukaydin Z, Guzel K. The Effect of Showing Images of the Foetus with the Virtual Reality Glass During Labour Process on Labour Pain, Birth Perception and Anxiety. J Clin Nurs. 2021 Aug;30(15-16):2301-2308. doi: 10.1111/jocn.15768. Epub 2021 May 6. PMID 33960065